CLINICAL TRIAL: NCT03953326
Title: Digital Intervention to Promote Physical Activity and Improve Cardiovascular Health Among Cancer Survivors
Brief Title: HeartPhone Cancer Survivors Trial 2019
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Futility in recruitment
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David E Conroy, Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00011271
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Leukemia; Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Leukemia; Lymphoma | interventions — Acetylcholine; Nitroprusside; Tosylarginine Methyl Ester

STUDY DESIGN:
Intervention Model Description: Single-group pre-post change
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HeartPhone Intervention (Experimental): Participants install the HeartPhone app on their smartphone. This app presents an image on a splash screen every time they activate their device. The image is randomly drawn from an image bank in the app. Repeated exposure to the image is designed to condition a more favorable automatic affective evaluation of physical activity and lead to increased physical activity.
  Interventions: Behavioral: HeartPhone app; Drug: Acetylcholine; Drug: Sodium Nitroprusside; Drug: L-Arginine, N2-((4-Methylphenyl)Sulfonyl)-, Methyl Ester

INTERVENTIONS:
Behavioral: HeartPhone app — Evaluative conditioning (temporally distributed micro-doses presented upon activation of smartphone screen)
Drug: Acetylcholine — Endothelium-dependent vasodilation is tested with the localized delivery of the neurotransmitter
Drug: Sodium Nitroprusside — Endothelium-independent vasodilation is tested with the localized delivery of the nitric oxide donor
Drug: L-Arginine, N2-((4-Methylphenyl)Sulfonyl)-, Methyl Ester — This nitric oxide inhibitor is continuously given during the localized delivery of the endothelium-dependent agonist acetycholine.

SUMMARY:
This is a behavioral study that will examine changes in physical activity and vascular health in response to a digital tool (app) that will appear on participant's lock screen of their Android phone. Participants will be asked to use this app for 3 months and to wear a Fitbit device continuously throughout the study. Participants will be asked to complete questionnaires, participate in fitness testing and measures of cardiovascular health at 3 months and 6 months after baseline assessments. The hypothesis is that exposure to the app will lead to increased physical activity volume and improved microvessel function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of breast cancer, leukemia, or lymphoma <15 yrs
* Completed chemotherapy with cardiotoxic anthracycline-based agents 1+ year ago
* English-proficiency
* Own & use smartphone with Android operating system

Main Study and Ancillary Study Exclusion Criteria:

* Currently receiving curative treatment for cancer
* 90+ min/week moderate (or greater) intensity PA
* Any medical contraindications on the Physical Activity Readiness Questionnaire
* Require an assistive device for mobility or has any other condition that may limit or prevent participation in moderate-intensity physical activity
* Current smoker
* Pregnant or planning to become pregnant in the next 6 mos/breastfeeding
* Allergy to test substances
* Allergy to latex

Ancillary Study:

* Taking metformin
* Current medications that could conceivably alter the cardiovascular or thermoregulatory control or responses (e.g. beta blockers, calcium channel blockers, angiotensin receptor blockers)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Physical activity volume | 3 month
  Daily step counts over 1-week from Fitbit device

SECONDARY OUTCOMES:
Microvessel function | 3 month
  Skin blood flow during perfusion of endothelium-dependent and independent agonists

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03953326/Prot_SAP_000.pdf